CLINICAL TRIAL: NCT01950299
Title: Interleukin-1 Blockade With Anakinra in Patients With ST-segment Elevation Myocardial Infarction - the Virginia Commonwealth University Anakinra Remodeling Trial 3
Brief Title: Interleukin-1 (IL-1) Blockade in Acute Myocardial Infarction (VCU-ART3)
Acronym: VCU-ART3
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20000024; 1R34HL121402-01 (NIH)
Record Dates: First submitted 2013-09-04; First posted 2013-09-25 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Anakinra (standard dose) (Experimental): Anakinra 100 mg daily for 14 days
  Interventions: Drug: Anakinra 100 mg; Drug: Placebo
- Anakinra (high dose) (Experimental): Anakinra 100 mg twice daily for 14 days
  Interventions: Drug: Anakinra 100 mg
- Placebo (Placebo Comparator): Placebo for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra 100 mg — Anakinra 100 mg starting immediately and then every 24 hours
  Other Names: Kineret
  Arms: Anakinra (high dose); Anakinra (standard dose)
Drug: Anakinra 100 mg — Anakinra 100 mg starting 12 hours after first dose and then every 24 hours (so that Anakinra is given every 12 hours)
  Other Names: Kineret
  Arms: Anakinra (high dose)
Drug: Placebo — Placebo 0.67 ml injections twice daily
  Other Names: Placebo injections twice daily
  Arms: Anakinra (standard dose); Placebo

SUMMARY:
VCU-ART3 is a double-blind randomized clinical trial of anakinra high dose vs anakinra standard dose vs placebo in patients with ST-segment elevation myocardial infarction (STEMI) measuring the effects on the acute rise and fall of the plasma C reactive protein levels during the first 14 days.

DETAILED DESCRIPTION:
VCU-ART3 is a double-blind randomized clinical trial of anakinra high dose vs anakinra standard dose vs placebo in patients with ST-segment elevation myocardial infarction (STEMI) measuring the effects on the acute rise and fall of the plasma C reactive protein levels during the first 14 days

ELIGIBILITY:
INCLUSION CRITERIA:

In order to be eligible for this study, patients must meet ALL the 3 Inclusion criteria and NONE of the Exclusion criteria.

1. Acute STEMI defined as chest pain (or equivalent) with an onset within 12 hours and ECG evidence of ST segment elevation (>1 mm) in 2 or more anatomically contiguous leads that is new or presumably new
2. Planned or completed coronary angiogram for potential intervention
3. Age>21

EXCLUSION CRITERIA:

* Inability to give informed consent
* Pregnancy
* Preexisting congestive heart failure (American Heart Association/American College of Cardiology class C-D, New York Heart Association III-IV)
* Preexisting severe left ventricular dysfunction (EF<20%)
* Preexisting severe valvular heart disease
* Active infections (acute or chronic) - excluding Hepatitis C Virus (HCV)+ with undetectable RNA
* Recent (<14 days) or active use of anti-inflammatory drugs (not including non-steroidal anti-inflammatory drugs [NSAIDs] or corticosteroids used for IV dye allergy only)
* Chronic inflammatory disease (including but not limited to rheumatoid arthritis, systemic lupus erythematosus)
* Active malignancy - excluding carcinoma in situ [any organ] and non-melanoma skin cancer
* Anticipated need for cardiac surgery
* Neutropenia (absolute neutrophil count<1,800/mm3)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2018-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Silvis MJM, Demkes EJ, Fiolet ATL, Dekker M, Bosch L, van Hout GPJ, Timmers L, de Kleijn DPV. Immunomodulation of the NLRP3 Inflammasome in Atherosclerosis, Coronary Artery Disease, and Acute Myocardial Infarction. J Cardiovasc Transl Res. 2021 Feb;14(1):23-34. doi: 10.1007/s12265-020-10049-w. Epub 2020 Jul 9. PMID 32648087
- [Derived] Abbate A, Trankle CR, Buckley LF, Lipinski MJ, Appleton D, Kadariya D, Canada JM, Carbone S, Roberts CS, Abouzaki N, Melchior R, Christopher S, Turlington J, Mueller G, Garnett J, Thomas C, Markley R, Wohlford GF, Puckett L, Medina de Chazal H, Chiabrando JG, Bressi E, Del Buono MG, Schatz A, Vo C, Dixon DL, Biondi-Zoccai GG, Kontos MC, Van Tassell BW. Interleukin-1 Blockade Inhibits the Acute Inflammatory Response in Patients With ST-Segment-Elevation Myocardial Infarction. J Am Heart Assoc. 2020 Mar 3;9(5):e014941. doi: 10.1161/JAHA.119.014941. Epub 2020 Mar 3. PMID 32122219
- [Derived] Van Tassell BW, Lipinski MJ, Appleton D, Roberts CS, Kontos MC, Abouzaki N, Melchior R, Mueller G, Garnett J, Canada J, Carbone S, Buckley LF, Wohlford G, Kadariya D, Trankle CR, Oddi Erdle C, Sculthorpe R, Puckett L, DeWilde C, Shah K, Angiolillo DJ, Vetrovec G, Biondi-Zoccai G, Arena R, Abbate A. Rationale and design of the Virginia Commonwealth University-Anakinra Remodeling Trial-3 (VCU-ART3): A randomized, placebo-controlled, double-blinded, multicenter study. Clin Cardiol. 2018 Aug;41(8):1004-1008. doi: 10.1002/clc.22988. Epub 2018 Aug 17. PMID 30033595

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra (Standard Dose) | Anakinra (High Dose) | Placebo
Started | 33 | 31 | 35
Completed | 22 | 27 | 28
Not Completed | 11 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra (Standard Dose) | Anakinra (High Dose) | Placebo | Total
Number analyzed (Participants) | 33 | 31 | 35 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 26 | 26 | 80
  >=65 years | 5 | 5 | 9 | 19
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [49 to 62] | 55 [45 to 61] | 56 [51 to 65] | 55 [49 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 5 | 19
  Male | 24 | 26 | 30 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 9 | 6 | 27
  White | 21 | 22 | 29 | 72
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 31 | 35 | 99

OUTCOME MEASURES:

1. Primary Outcome: Acute Phase Response (CRP Levels)
Description: Comparison of area-under-the-curve for CRP up to day 14
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: mg x day/L (milligram x day/liter)
Arm/Group | Anakinra (Standard Dose) | Anakinra (High Dose) | Placebo
Number analyzed (Participants) | 22 | 27 | 28
mg x day/L (milligram x day/liter) | 60.03 [23.50 to 138.72] | 86.35 [43.44 to 122.73] | 213.75 [131.36 to 394.20]

2. Secondary Outcome: Left Ventricular End-systolic Volume
Description: Placebo corrected interval change in left ventricular end-systolic volume over 12 months
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: mL (milliliters)
Arm/Group | Anakinra (Standard Dose) | Anakinra (High Dose) | Placebo
Number analyzed (Participants) | 20 | 21 | 25
mL (milliliters) | 0 [-8 to 6] | 4 [-14 to 11] | -4 [-15 to 1]

3. Secondary Outcome: Left Ventricular Ejection Fraction
Description: Placebo-corrected interval changes in left ventricular ejection fraction over 12 months
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: % (Left ventricular ejection fraction)
Arm/Group | Anakinra (Standard Dose) | Anakinra (High Dose) | Placebo
Number analyzed (Participants) | 20 | 21 | 25
% (Left ventricular ejection fraction) | 4 [-2 to 7] | 5 [-1 to 5] | 3 [-2 to 9]

4. Secondary Outcome: Heart Failure
Description: New onset of heart failure symptoms (NYHA II-IV)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra (Standard Dose) | Anakinra (High Dose) | Placebo
Number analyzed (Participants) | 33 | 31 | 35
Participants | 3 | 3 | 9

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Anakinra (Standard Dose) | Anakinra (High Dose) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31 | 1/35
Serious Adverse Events (participants affected / at risk) | 6/33 | 7/31 | 8/35
Other Adverse Events (participants affected / at risk) | 6/33 | 8/31 | 1/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (Standard Dose) (N=33) | Anakinra (High Dose) (N=31) | Placebo (N=35)
Death (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Heart Failure Hospitalization (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 3 (3) | 6 (6) | 5 (5)
Unstable Angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Revascularization (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Stroke/Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (Standard Dose) (N=33) | Anakinra (High Dose) (N=31) | Placebo (N=35)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT01950299/Prot_SAP_000.pdf